CLINICAL TRIAL: NCT01483222
Title: Comparison of Inelastic and Elastic Lumbosacral Orthoses on Low Back Pain Prevention in Hospital Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Hongbin Lu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20101201
Record Dates: First submitted 2011-11-26; First posted 2011-12-01 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Braces; Prevention
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- QUIKDRAW Pro (Experimental): Wearing an inelastic lumbar support for 6 months
  Interventions: Device: QUIKDRAW Pro, Aspen Medical Products
- MUELLER 4581 (Experimental): Wearing an elastic lumbar support for 6 months
  Interventions: Device: MUELLER 4581, Mueller Sports Medicine
- Blank Control (No Intervention): Receiving no intervention

INTERVENTIONS:
Device: QUIKDRAW Pro, Aspen Medical Products — Wearing an inelastic lumbar support (QUIKDRAW Pro, Aspen Medical Products) for 6 months
  Other Names: Lumbar belt, Lumbar orthoses, Lumbar brace
  Arms: QUIKDRAW Pro
Device: MUELLER 4581, Mueller Sports Medicine — Wearing an elastic lumbar support (MUELLER 4581, Mueller Sports Medicine) for 6 months
  Other Names: Lumbar belt, Lumbar orthoses, Lumbar brace
  Arms: MUELLER 4581

SUMMARY:
The main objective of this study is to investigate the efficacy of two different design characteristics of lumbar support for low back pain prevention in hospital nurses.

DETAILED DESCRIPTION:
Low back pain occurs frequently and is one of the most costly health problems affecting industry and society. Prevention of low back pain is important both for the individual patient and from an economic perspective. Therefore, there are many measures available that claim to reduce low back pain and its recurrence. The most commonly used preventive strategies are fitness exercises, lumbar supports, education on back mechanics and lifting techniques, and ergonomic adjustments. However, their efficacy is still uncertain. The main objective of this study is to investigate the efficacy of two different design characteristics of lumbar support for low back pain prevention in hospital nurses. Investigators hope that those two types of lumbar support will reduce the incidence of low back pain and sick leave days. In addition, Investigators hypothesize that there are some differences on outcome measures between those two types of lumbar support. Enrolled subjects will be randomly assigned to one of the following three groups. The first group will wear an inelastic lumbar support for 6 months. The second group will wear an elastic lumbar support for 6 months. The third group will receive no intervention. After the completion of 6-month intervention, a further 6 months fellow-up will be added.

ELIGIBILITY:
Inclusion Criteria:

1. Female between 20 and 25 years of age
2. Subjects who have worked as a nurse less than two years and will continue working as a nurse no less than one year
3. Job contents including moving and lifting patients, long-time standing and frequent bending
4. Subjects who do not participate any other study concerning pain prevention currently and in the next year

Exclusion Criteria:

1. Subjects who are experiencing low back pain symptoms at the time of inquiry, regardless of acute or chronic, and seeking medical care currently
2. Subjects who have experienced 2 or more episodes (on 2 consecutive days) of low back pain symptoms in the 12 months before the inquiry
3. Subjects who are suffering from any other chronic pain disorders symptomatically
4. Subjects who have used a lumbar support during the last 6 months
5. Subjects with specific low back pain (like infection, tumors, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome or cauda equina syndrome, spinal stenosis or spondylolysis)
6. Subjects who have had a spinal operation
7. Subjects who are suffering from chronic cardiac, respiratory, liver and kidney complaint symptomatically
8. Subjects who are suffering from diseases that might be aggravated by increased intra-abdominal pressure, like hernia
9. Subjects who are suffering from chronic gastrointestinal disorders symptomatically
10. Subjects who are pregnant, planning to have a baby in 1 year or less than 6 months after delivery
11. Subjects who are suffering from serious somatic disease and/or psychic disease

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The incidences of low back pain | 12 months after initiation
The sick leave days due to low back pain | 12 months after initiation

SECONDARY OUTCOMES:
Medical care utilization | 12 months after initiation
Adverse Effects | 12 months after initiation
Quality of life | 12 months after initiation

CONTACTS AND LOCATIONS:
Overall Officials: Hongbin Lu, M.D. & Ph.D., Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China